CLINICAL TRIAL: NCT00555659
Title: Prospective Clinical Evaluation of the New Aegis Plate for Anterior Interbody
Brief Title: Prospective Clinical Evaluation of the New Aegis Plate for Anterior Interbody Fusions
Acronym: Aegis
Status: Completed | Type: Observational
Sponsor: Columbia Orthopaedic Group, LLP (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Principal Investigator, John Miles, MD, Investigator, Columbia Orthopaedic Group, LLP
Other Study IDs: 1094241
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Degeneration; Spondylosis; Spondylolithesis; Stenosis
Keywords: Degeneration; Spondylosis; Spondylolisthesis; Stenosis
MeSH Terms: conditions — Spondylosis; Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction: Degenerative changes of the discs and facet joints in the lumbar spine can result in pain and disability from spondylosis, spondylolisthesis and stenosis. Patients who are suffering with back and/or leg pain are potential candidates for an ALIF procedure.

Purpose: To assess and compare clinical outcomes and fusion rates in patients undergoing an instrumented ALIF procedure. Comparisons in all variables will be made across diagnostic categories. Comparisons between type of interbody spacer, graft type, and type of instrumentation will also be made

DETAILED DESCRIPTION:
To assess and compare clinical outcomes and fusion rates in patients undergoing an instrumented ALIF procedure. Comparisons in all variables will be made across diagnostic categories. Comparisons between type of interbody spacer, graft type, and type of instrumentation will also be made.

This study is part of a larger Continuous Quality Improvement initiative at the Columbia Orthopaedic Group. The purpose of this effort is to improve surgical and non-surgical outcomes by using rigorous statistical analysis of our outcomes to guide our treatment decisions. Through an iterative feedback process we hope to optimize patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Standard of care

Exclusion Criteria:

* Standard of care

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person who comes into the clinic and gives consent to participate in this prospective study.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2007-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Intake data will include all fields traditionally associated with a detailed note. Subsequent visit instruments will include visual analog scale and oswestry disability index. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John D Miles, MD, Principal Investigator — Columbia Orthopaedic Group, LLP
Locations (1):
- Columbia Orthopaedic Group, Columbia, Missouri, United States